CLINICAL TRIAL: NCT01186913
Title: A Prospective Natural History Study of Diagnosis, Treatment and Outcomes of Children With SCID Disorders (RDCRN PIDTC-6901)
Brief Title: Natural History Study of SCID Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Primary Immune Deficiency Treatment Consortium (PIDTC) (Other); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT RDCRN PIDTC-6901; NCT02108067 (obsolete NCT alias)
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Severe Combined Immunodeficiency (SCID); Leaky SCID; Omenn Syndrome; Reticular Dysgenesis; ADA SCID; XSCID
Keywords: Severe Combined Immunodeficiency (SCID); natural history study; SCID treatment
MeSH Terms: conditions — Severe Combined Immunodeficiency; Reticular dysgenesis; Severe combined immunodeficiency due to adenosine deaminase deficiency; X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples, tissue, and bone marrow samples collected during participation in this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Stratum A: Typical SCID +HCT: Stratum A: Typical Severe Combined Immunodeficiency (SCID) treated with HCT therapy.
  Participants with typical (formerly referred to as classic) SCID + allogeneic hematopoietic stem cell transplantation (HCT) therapy according to standard of care, per local protocol.
- Stratum B: Atypical SCID +HCT: Stratum B: Atypical Severe Combined Immunodeficiency (SCID) treated with HCT therapy.
  Participants with leaky SCID, Omenn syndrome, or Reticular Dysgenesis (RS) + allogeneic hematopoietic stem cell transplantation (HCT) therapy according to standard of care, per local protocol.
- Stratum C:SCID +Non-HCT: Stratum C: Severe Combined Immunodeficiency (SCID) who receive alternative therapy per standard of care, non-standard care and/or investigational. This stratum includes:
  * Adenosine Deaminase-Deficient SCID (ADA Deficient SCID) with intention to treat with Polyethylene Glycol -Adenosine Deaminase Enzyme Replacement Therapy (PEG-ADA ERT)
  * ADA Deficient SCID with intention to treat with gene therapy
  * X-linked SCID (XSCID) with intention to treat with gene therapy
  * Any individual with SCID previously treated with a thymus transplant (includes intention to treat with HCT, as well as PEG-ADA ERT or gene therapy)

SUMMARY:
This study is a prospective evaluation of children with Severe Combined Immune Deficiency (SCID) who are treated under a variety of protocols used by participating institutions. In order to determine the patient, recipient and transplant-related variables that are most important in determining outcome, study investigators will uniformly collect pre-, post- and peri-transplant (or other treatment) information on all children enrolled into this study.

Children will be divided into three strata:

* Stratum A: Typical SCID with virtual absence of autologous T cells and poor T cell function
* Stratum B: Atypical SCID (leaky SCID, Omenn syndrome and reticular dysgenesis with limited T cell diversity or number and reduced function), and
* Stratum C: ADA deficient SCID and XSCID patients receiving alternative therapy including PEG-ADA ERT or gene therapy.

Each Group/Cohort Stratum will be analyzed separately.

DETAILED DESCRIPTION:
This study follows participants with SCID prospectively, meaning the study enrolls participants where there is a plan to receive a blood and marrow transplant, enzyme therapy, or gene therapy in the future. Participants are then followed according to a schedule set out by the study protocol after the procedure. There are no experimental therapies on this study.

The goal of this study is to learn more about: (1) outcomes from the treatment of SCID in the modern era of medicine (2) what factors lead to the best long-term outcomes, such as best donor, conditioning regimen, timing of transplant, etc., and (3) what impact newborn screening and the early diagnosis of SCID has had on the long-term outcomes following BMT or gene therapy. Information is also being gathered on how and when the immune system recovers after bone marrow transplant (BMT), quality of life for long-term survivors, and about whether children develop normally after treatment.

This natural history study is the largest coordinated prospective study of participants with SCID ever performed. Information that investigators will learn, both now and in the future, will help doctors and other health professionals to better treat children with SCID.

ELIGIBILITY:
Inclusion Criteria:

Stratum A: Typical SCID (formerly referred to as Classic SCID)- -Subjects who meet the following inclusion criteria and the intention is to treat with allogeneic hematopoietic cell transplant (HCT) are eligible for enrollment into Stratum A (Typical SCID) of the study:

* Absence or very low number of T cells (CD3 T cells <300/microliter) AND
* No or very low T cell function (<10% of lower limit of normal) as measured by response to phytohemagglutinin (PHA) OR
* T cells of maternal origin present.

Stratum B: Leaky SCID, Omenn Syndrome, Reticular Dysgenesis-

-Subjects who meet the following criteria and the intention is to treat with HCT are eligible for enrollment into Stratum B:

Leaky SCID:

* Maternal lymphocytes tested for and not detected AND
* Either one or both of the following (a,b) :

  * a.) <50% of lower limit of normal T cell function as measured by response to PHA, OR response to anti-CD3/CD28 antibody
  * b.) Absent or <30% of lower limit of normal proliferative responses to candida and tetanus toxoid antigens
* AND at least two of the following (a through e):

  * a.) Reduced number of CD3 T cells

    * age ≤2 years: <1500/microliter
    * age >2 years and ≤4 years: <800/microliter
    * age >4 years: <600/microliter
  * b.) ≥80% of CD3+ or CD4+ T cells that are CD45RO+

    * AND/OR >80% of CD3+ or CD4+ T cells are CD62L negative
    * AND/OR >50% of CD3+ or CD4+T cells express HLA-DR (at <4 years of age)
    * AND/OR are oligoclonal T cells
  * c.) Hypomorphic mutation in IL2RG in a male, or homozygous hypomorphic mutation or compound heterozygosity with ≥1 hypomorphic mutation in an autosomal SCID-causing gene
  * d.) Low T Cell Receptor Excision Circles (TRECs) and/or the percentage of CD4+/45RA+/CD31+ or CD4+/45RA+/CD62L+ cells is below the lower limit of normal.
  * e.) Functional testing in vitro supporting impaired, but not absent, activity of the mutant protein, AND
* Does not meet criteria for Omenn Syndrome.

Omenn Syndrome:

* Generalized skin rash
* Maternal lymphocytes tested for and not detected;

  --Note: If maternal engraftment was not assessed and ruled out, the subject is not eligible as Omenn Syndrome.
* ≥80% of CD3+ or CD4+ T cells are CD45RO+ AND/OR

  * 80% of CD3+ or CD4+T cells are CD62L negative AND/OR
  * 50% of CD3+ or CD4+ T cells express HLA-DR (at <2 years of age);
* Absent or low (< 30% lower limit of normal) T cell proliferation response to antigens (Candida, tetanus) to which the subject has been exposed

NOTE: If proliferation to antigen was not performed, but at least 4 of the following 9 supportive criteria, at least one of which must be among those marked with an asterisk (*) below are present, the subject is eligible as Omenn Syndrome:

* Hepatomegaly
* Splenomegaly
* Lymphadenopathy
* Elevated IgE
* Elevated absolute eosinophil count
* *Oligoclonal T cells measured by CDR3 length or flow cytometry
* *Proliferation to PHA is reduced <50% of lower limit of normal or SI <30
* *Hypomorphic mutation in a SCID causing gene
* Low TRECS and/or the percentage of CD4+/45RA+/CD31+ or CD4+/45RA+/CD62L+ cells is below the lower limit of normal.

Reticular Dysgenesis:

* Absence or very low number of T cells (CD3 <300/µL
* No or very low (<10% lower limit of normal) T cell response to PHA
* Severe neutropenia (absolute neutrophil count < 200 /µL) AND
* ≥2 of the following (a,b,c):

  * a.) Sensori-neural deafness
  * b.) Deficiency of marrow granulopoiesis on bone marrow examination
  * c.) A pathogenic mutation in the adenylate kinase 2 (AK2) gene identified.

Stratum C:

Subjects who meet the following criteria and the intention is to treat with therapy other than allogeneic HCT, primarily PEG-ADA ERT or gene therapy with autologous modified (gene transduced) cells, are eligible for enrollment into

Stratum C:

* ADA Deficient SCID with intention to treat with PEG-ADA ERT
* ADA Deficient SCID with intention to treat with gene therapy
* X-linked SCID with intention to treat with gene therapy
* Any SCID patient previously treated with a thymus transplant (includes intention to treat with HCT, as well as PEG-ADA ERT or gene therapy)
* Any SCID patient who received therapy for SCID deemed "non-standard" or "investigational", including in utero procedures.

Exclusion Criteria:

-Subjects who meet any of the following exclusion criteria are disqualified from enrollment in Strata A, B, or C of the study:

* Presence of an Human Immunodeficiency Virus (HIV) infection (by PCR) or other cause of secondary immunodeficiency
* Presence of DiGeorge syndrome
* MHC Class I and MHC Class II antigen deficiency, and
* Metabolic conditions that imitate SCID or related disorders such as folate transporter deficiency, severe zinc deficiency or transcobalamin deficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with SCID spectrum disorders that have undergone diagnostic workup per local center practice and referred for enrollment in this natural history study at one of the participating institutions (clinical research site locations).
Sampling Method: Non-Probability Sample
Enrollment: 690 (Estimated)
Dates: Start 2010-09-02 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) at Month 6 Post HCT | Month 6 Post HCT
  Assess the overall survival (OS) for participants after hematopoietic stem cell transplantation (HCT) for treatment of Severe Combined Immunodeficiency (SCID).
  The time to this event is the time from HCT to death or last follow-up (whichever occurs first). All participants will be followed for a minimum of 6 months from HCT. Overall survival will be estimated at 6 months.
Overall Survival (OS) at Year 2 Post HCT | Year 2 Post HCT
  Assess the overall survival (OS) for participants after hematopoietic stem cell transplantation (HCT) for treatment of Severe Combined Immunodeficiency (SCID).
  The time to this event is the time from HCT to death or last follow-up (whichever occurs first). All participants will be followed for a minimum of 6 months from HCT. Overall survival will be estimated at 2 years.
Overall Survival (OS) at Year 5 Post HCT | Year 5 Post HCT
  Assess the overall survival (OS) for participants after hematopoietic stem cell transplantation (HCT) for treatment of Severe Combined Immunodeficiency (SCID).
  The time to this event is the time from HCT to death or last follow-up (whichever occurs first). All participants will be followed for a minimum of 6 months from HCT. Overall survival will be estimated at 5 years.
Overall Survival (OS) at Year 8 Post HCT | Year 8 Post HCT
  Assess the overall survival (OS) for participants after hematopoietic stem cell transplantation (HCT) for treatment of Severe Combined Immunodeficiency (SCID).
  The time to this event is the time from HCT to death or last follow-up (whichever occurs first). All participants will be followed for a minimum of 6 months from HCT. Overall survival will be estimated at 8 years.

SECONDARY OUTCOMES:
T Cell Reconstitution by Stratum-Month 6, Year 2, Year 5 and Year 8 Post-SCID Treatment | From SCID Treatment (HCT, ERT or GT) to Month 6, Year 2, Year 5 and Year 8 Post-SCID Treatment
  A measure of immune reconstitution defined by the presence of three out of four of:
  1. Lymphocyte proliferation to PHA ≥50% of lower limit of normal control
  2. Total CD3+ > 1000 / microliter
  3. Total CD4+ > 500 / microliter
  4. Total CD4+ CD45RA+ > 200 / microliter
  AND, for participants who received allogeneic HCT:
  -Donor T cell chimerism ≥80%
B Cell Reconstitution by Stratum-Month 6, Year 2, Year 5 and Year 8 Post-SCID Treatment | From SCID Treatment (HCT, ERT or GT) to Month 6, Year 2, Year 5 and Year 8 Post-SCID Treatment
  A measure of immune reconstitution defined by:
  -Intravenous Immunoglobulin (IVIG) independence and at least three of the following:
  1. Normal IgA and IgM levels for age
  2. Normal IgG levels for age, independent of supplemental gammaglobulin
  3. Isohemagglutinins ≥1:8
  4. Specific antibody production while off IVIG
Engraftment at Day 100, Month 6, Year 2, Year 5 and Year 8 Post-HCT | From HCT to Month 6, Year 2, Year 5 and Year 8 Post-HCT
  Whole-blood engraftment and engraftment in T-, B-, or Natural Killer (NK)-cell subsets will be assessed.
  For whole blood and subsets*, the following engraftment criteria will be used:
  * < 5% donor = autologous reconstitution
  * 5-80% donor = mixed chimerism
  * ≥ 80% donor = full chimerism
    * Subsets:
      * CD3
      * CD19
      * CD14 and/or CD15 (myeloid cells)
      * CD3- CD56+ NK cells
  Outcome analysis restricted to participants with hematopoietic (stem) cell transplantation (HCT) intervention.
Time to Resolution of Infections Diagnosed Prior to HCT | Through study completion, up to 8 years post-HCT
  Time to resolution of any "pre-HCT" infections-bacterial, viral or fungal. Participants who are alive without resolving their pre-HCT infections will be considered censored at last contact.
  Resolution of pre-existing infection defined by:
  * Participant being clinically well,
  * Participant off treatment for infection(s), and/or
  * Negative culture/PCR assay.
  Outcome analysis restricted to participants with pre-hematopoietic (stem) cell transplantation (HCT) opportunistic infections.
Incidence of New Infections Post-HCT | From HCT to Day 100, Month 6, Year 1, Year 2, Year 5, and Year 8 post-HCT
  The occurrence of new documented bacterial, viral, or fungal infections-by site of disease, organism, date of onset, and resolution- post-HCT.
  Participants who are alive without infection will be considered censored at last contact.
  Outcome analysis restricted to participants with hematopoietic (stem) cell transplantation (HCT).
Proportion of Participants Achieving Normal Nutritional Status Post-HCT | Baseline (Pre-HCT) to Year 1, Year 2, Year 5 and Year 8 Post-HCT
  Normal nutrition status defined by:
  * Absence of chronic diarrhea and/or
  * No longer requiring supplemental nutrition (i.e., tube feeding or TPN).
    * TPN: total parenteral nutrition
  Outcome analysis restricted to participants with hematopoietic (stem) cell transplantation (HCT) intervention.
Longitudinal Analysis: Growth Percentile in Body Height | Baseline (Pre-HCT), Year 1, Year 2, Year 5 and Year 8 Post-HCT
  Participant's height will be superimposed against gender specific standard growth charts.
Longitudinal Analysis: Growth Percentile in Body Weight | Baseline (Pre-HCT), Year 1, Year 2, Year 5 and Year 8 Post-HCT
  Participant's weight will be superimposed against gender specific standard growth charts.
Incidence of Acute Graft Versus Host Disease (GVHD) Post-HCT | From HCT to Day 100 and Month 6 post-HCT
  Occurrence of acute GVHD. Any skin, gastrointestinal or liver abnormalities fulfilling the consensus criteria of Grades II-IV acute GVHD or grades III-IV acute GVHD are considered events.
  Participants alive without acute GVHD will be censored at the time of last follow-up.
  Outcome analysis restricted to participants with hematopoietic (stem) cell transplantation (HCT) intervention.
Incidence of Chronic Graft Versus Host Disease (GVHD) Post-HCT | From HCT to Month 6, Year 1,Year 2, Year 5 and Year 8 Post-HCT
  Occurrence of chronic GVHD in any organ system fulfilling the criteria of limited or extensive chronic GVHD. Participants alive without chronic GVHD will be censored at time of last follow-up.
  Outcome analysis restricted to participants with hematopoietic (stem) cell transplantation (HCT).
Incidence of Autoimmunity Requiring Treatment by Stratum- Month 6, Year 2, Year 5 and Year 8 Post-SCID Treatment | From SCID Treatment (HCT, ERT or GT) to Month 6, Year 2, Year 5 and Year 8 Post-SCID Treatment
  Occurrence of autoimmunity requiring treatment with immunosuppression or other therapy. Participants alive without autoimmunity will be censored at time of last follow-up.
  Date of onset and type of treatment will be collected on:
  * Autoimmune hypothyroidism
  * Autoimmune cytopenia (hemolytic anemia, thrombocytopenia, neutropenia)
  * Arthritis
  * Myositis
  * Nephritis
  * Bronchiolitis obliterans or other pulmonary autoimmune disease
  * Vitiligo
  * Alopecia
  * Inflammatory bowel disease
  * Neurodegeneration
  * Vasculitis
Infant Neurocognitive Development By Stratum Measured by Bayley's Scales for Infant Development 3rd edition (BSID-III-R) | Baseline (Pre-SCID Treatment-HCT, ERT or GT),Year 1, Year 2, Year 4, Year 5 and Year 8 Post-SCID Treatment
  Infant development as measured by Bayley's scales for infant development 3rd edition (BSID-III-R, Bayley, 2006).] The BSID III-R is a standardized developmental exam that is normalized to the age of the child in months. The mean adjusted score is 100 with a standard deviation of 15 (higher being better). Evaluation conducted as per standard of care in participants ≤30 months of age.
Neurocognitive Development By Stratum Measured by Vineland Adaptive Behavior Scales, Second Edition (Vineland II) | Baseline (Pre-SCID Treatment-HCT, ERT or GT),Year 1, Year 2, Year 4, Year 5 and Year 8 Post-SCID Treatment
  The Vineland II measures the personal and social skills of individuals from birth through adulthood. Since adaptive behavior refers to an individual's typical performance of the day-to-day activities required for personal and social sufficiency, these scales assess what a person actually does, rather than what he or she is able to do.
  Summary: The Vineland II is a measure of adaptive behavior in children, adolescents and adults. It yields an overall standard score (Adaptive Behavior Composite, ABC) and age standard scores in four domains: Communication, Daily Living Skills, Motor Skills, and Maladaptive Behaviour Index.
  ABC scores have a mean of 100 and a standard deviation of 15 (range = 20 to 160). Higher scores suggest a higher level of adaptive functioning. A rise in standard scores from Baseline indicates improvement.
  Evaluation as per standard of care.
Neurocognitive Development By Stratum Measured by Wechsler Preschool and Primary Intelligence Scale of Intelligence, Third Edition (WPPSI III) | Baseline (Pre-SCID Treatment-HCT, ERT or GT),Year 1, Year 2, Year 4, Year 5 and Year 8 Post-SCID Treatment
  Cognitive ability assessed using the WPPSI III. The WPPSI-III has been developed and standardized for children ages 2 years, 6 months through 7 years, 3 months of age. The WPPSI-III yields a Verbal Score, a Performance Score, a General Language Score, and a Full Scale Score. These scores have a mean of 100 and a standard deviation of 15. The range of possible values is 50 (worst value) to 150 (best value).
  Evaluation as per standard of care.
Neurocognitive Assessment by Stratum Using the Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) | Baseline (Pre-SCID Treatment-HCT, ERT or GT),Year 1, Year 2, Year 4, Year 5 and Year 8 Post-SCID Treatment
  The WISC-IV is designed for children 6 years 0 months to 16 years 11 months. The Full Scale IQ, ranges from 45 to 155 with a mean of 100 and standard deviation of 15. Higher scores indicate stronger cognitive function. Scores between 90 and 110 are considered to be within the range of average IQ. Evaluation in accordance with standard of care, participant ages 6 years and above.
Incidence of Complications of HCT Requiring Treatment | From HCT to Month 6, Year 1,Year 2, Year 5 and Year 8 Post-HCT
  Occurrence of health event(s) classified as an HCT treatment complication, including but not limited to:
  * Veno-occlusive disease
  * Thrombotic thrombocytopenic purpura
  * Bronchiolitis obliterans / chronic lung disease
  * Seizures
  * Hypertension
  Outcome analysis restricted to participants with hematopoietic (stem) cell transplantation (HCT) intervention.
Comparison of Quality of Life (QOL) By Stratum Prior to and After SCID Treatment: Scores for Pediatric Quality of Life Questionnaire (Peds-QL) | Baseline (Pre-SCID Treatment-HCT, ERT or GT) to Year 1, Year 2, Year 4, Year 5 and Year 8 Post-SCID Treatment
  The Peds-QL is a generic Health-Related Quality of Life (HR QoL) instrument designed specifically for a pediatric population. It captures the following domains: general health/activities, feelings/emotional, social functioning, school functioning. Higher scores indicate better quality of life (QOL) for all domains of the Peds-QL. This modular instrument uses a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. 4 dimensions (physical, emotional, social, & school functioning) are scored.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Dvorak, MD, Principal Investigator — UCSF Children's Hospital; Morton J. Cowan, MD, Principal Investigator — UCSF Children's Hospital
Locations (44):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California San Francisco Children's Hospital, San Francisco, California
  - Children's Hospital Denver, Denver, Colorado
  - Alfred I. duPont Hospital for Children/Nemours, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta/Emory University School of Medicine, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital/Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - NIH Clinical Center Genetic Immunotherapy Section, Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Hospital, Rochester, Minnesota
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University St Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center/ Golisano Children's Hospital, Rochester, New York
  - New York Medical College, Maria Fareri Children's Hospital, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals-Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center/Children's of Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Methodist Children's Hospital of South Texas/Texas Transplant Institute, San Antonio, Texas
  - Primary Children's Medical Center/University of Utah, Salt Lake City, Utah
  - Seattle Children's Research Institute, Seattle, Washington
  - University of Wisconsin/ American Family Children's Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Background] Griffith LM, Cowan MJ, Kohn DB, Notarangelo LD, Puck JM, Schultz KR, Buckley RH, Eapen M, Kamani NR, O'Reilly RJ, Parkman R, Roifman CM, Sullivan KE, Filipovich AH, Fleisher TA, Shearer WT. Allogeneic hematopoietic cell transplantation for primary immune deficiency diseases: current status and critical needs. J Allergy Clin Immunol. 2008 Dec;122(6):1087-96. doi: 10.1016/j.jaci.2008.09.045. Epub 2008 Nov 6. PMID 18992926
- [Result] Dvorak CC, Cowan MJ, Logan BR, Notarangelo LD, Griffith LM, Puck JM, Kohn DB, Shearer WT, O'Reilly RJ, Fleisher TA, Pai SY, Hanson IC, Pulsipher MA, Fuleihan R, Filipovich A, Goldman F, Kapoor N, Small T, Smith A, Chan KW, Cuvelier G, Heimall J, Knutsen A, Loechelt B, Moore T, Buckley RH. The natural history of children with severe combined immunodeficiency: baseline features of the first fifty patients of the primary immune deficiency treatment consortium prospective study 6901. J Clin Immunol. 2013 Oct;33(7):1156-64. doi: 10.1007/s10875-013-9917-y. Epub 2013 Jul 2. PMID 23818196
- [Result] Shearer WT, Dunn E, Notarangelo LD, Dvorak CC, Puck JM, Logan BR, Griffith LM, Kohn DB, O'Reilly RJ, Fleisher TA, Pai SY, Martinez CA, Buckley RH, Cowan MJ. Establishing diagnostic criteria for severe combined immunodeficiency disease (SCID), leaky SCID, and Omenn syndrome: the Primary Immune Deficiency Treatment Consortium experience. J Allergy Clin Immunol. 2014 Apr;133(4):1092-8. doi: 10.1016/j.jaci.2013.09.044. Epub 2013 Nov 28. PMID 24290292
- [Result] Haddad E, Allakhverdi Z, Griffith LM, Cowan MJ, Notarangelo LD. Survey on retransplantation criteria for patients with severe combined immunodeficiency. J Allergy Clin Immunol. 2014 Feb;133(2):597-9. doi: 10.1016/j.jaci.2013.10.022. Epub 2013 Dec 10. No abstract available. PMID 24331379
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Pai SY, Ballard B, Bauer SC, Bleesing JJ, Boyle M, Brower A, Buckley RH, van der Burg M, Burroughs LM, Candotti F, Cant AJ, Chatila T, Cunningham-Rundles C, Dinauer MC, Dvorak CC, Filipovich AH, Fleisher TA, Bobby Gaspar H, Gungor T, Haddad E, Hovermale E, Huang F, Hurley A, Hurley M, Iyengar S, Kang EM, Logan BR, Long-Boyle JR, Malech HL, McGhee SA, Modell F, Modell V, Ochs HD, O'Reilly RJ, Parkman R, Rawlings DJ, Routes JM, Shearer WT, Small TN, Smith H, Sullivan KE, Szabolcs P, Thrasher A, Torgerson TR, Veys P, Weinberg K, Zuniga-Pflucker JC; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) report. J Allergy Clin Immunol. 2014 Feb;133(2):335-47. doi: 10.1016/j.jaci.2013.07.052. Epub 2013 Oct 15. PMID 24139498
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Shearer WT, Burroughs LM, Torgerson TR, Decaluwe H, Haddad E; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) update. J Allergy Clin Immunol. 2016 Aug;138(2):375-85. doi: 10.1016/j.jaci.2016.01.051. Epub 2016 Apr 22. PMID 27262745
- [Result] Pai SY, Logan BR, Griffith LM, Buckley RH, Parrott RE, Dvorak CC, Kapoor N, Hanson IC, Filipovich AH, Jyonouchi S, Sullivan KE, Small TN, Burroughs L, Skoda-Smith S, Haight AE, Grizzle A, Pulsipher MA, Chan KW, Fuleihan RL, Haddad E, Loechelt B, Aquino VM, Gillio A, Davis J, Knutsen A, Smith AR, Moore TB, Schroeder ML, Goldman FD, Connelly JA, Porteus MH, Xiang Q, Shearer WT, Fleisher TA, Kohn DB, Puck JM, Notarangelo LD, Cowan MJ, O'Reilly RJ. Transplantation outcomes for severe combined immunodeficiency, 2000-2009. N Engl J Med. 2014 Jul 31;371(5):434-46. doi: 10.1056/NEJMoa1401177. PMID 25075835
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Puck JM, Buckley RH, Candotti F, Conley ME, Fleisher TA, Gaspar HB, Kohn DB, Ochs HD, O'Reilly RJ, Rizzo JD, Roifman CM, Small TN, Shearer WT; Workshop Participants. Improving cellular therapy for primary immune deficiency diseases: recognition, diagnosis, and management. J Allergy Clin Immunol. 2009 Dec;124(6):1152-60.e12. doi: 10.1016/j.jaci.2009.10.022. PMID 20004776
- [Result] Dvorak CC, Haddad E, Buckley RH, Cowan MJ, Logan B, Griffith LM, Kohn DB, Pai SY, Notarangelo L, Shearer W, Prockop S, Kapoor N, Heimall J, Chaudhury S, Shyr D, Chandra S, Cuvelier G, Moore T, Shenoy S, Goldman F, Smith AR, Sunkersett G, Vander Lugt M, Caywood E, Quigg T, Torgerson T, Chandrakasan S, Craddock J, Davila Saldana BJ, Gillio A, Shereck E, Aquino V, DeSantes K, Knutsen A, Thakar M, Yu L, Puck JM. The genetic landscape of severe combined immunodeficiency in the United States and Canada in the current era (2010-2018). J Allergy Clin Immunol. 2019 Jan;143(1):405-407. doi: 10.1016/j.jaci.2018.08.027. Epub 2018 Sep 5. PMID 30193840
- [Derived] Rayes A, Logan BR, Liu X, Dara J, Buckley RH, Oved JH, Kapoor N, Kapadia M, Chandra S, Martinez CA, Bunin N, Chandrakasan S, Chen K, Bednarski JJ, Haines HL, Eissa H, Talano JM, Keller MD, Ebens CL, Chaudhury S, Shereck EB, Aquino VM, Knutsen AP, Alexander JL, Gillio AP, Chellapandian D, Shah AJ, Miller HK, Vander Lugt MT, Seroogy CM, Dorsey MJ, Mousallem T, Parrott RE, O'Reilly RJ, Aguayo-Hiraldo PI, Prockop SE, Davila Saldana BJ, Thakar MS, Burroughs LM, Torgerson TR, Leiding JW, Marsh RA, Griffith LM, Pulsipher MA, Kohn DB, Notarangelo LD, Cowan MJ, Puck JM, Cuvelier GDE, Heimall J, Haddad E, Pai SY, Dvorak CC. Outcomes Following Matched Sibling Donor Transplantation for Severe Combined Immunodeficiency: A Report from the PIDTC. Blood Adv. 2025 Nov 25:bloodadvances.2025016812. doi: 10.1182/bloodadvances.2025016812. Online ahead of print. PMID 41289158
- [Derived] Cuvelier GDE, Logan BR, Prockop SE, Buckley RH, Kuo CY, Griffith LM, Liu X, Yip A, Hershfield MS, Ayoub PG, Moore TB, Dorsey MJ, O'Reilly RJ, Kapoor N, Pai SY, Kapadia M, Ebens CL, Forbes Satter LR, Burroughs LM, Petrovic A, Chellapandian D, Heimall J, Shyr DC, Rayes A, Bednarski JJ, Chandra S, Chandrakasan S, Gillio AP, Madden L, Quigg TC, Caywood EH, Davila Saldana BJ, DeSantes K, Eissa H, Goldman FD, Rozmus J, Shah AJ, Vander Lugt MT, Thakar MS, Parrott RE, Martinez C, Leiding JW, Torgerson TR, Pulsipher MA, Notarangelo LD, Cowan MJ, Dvorak CC, Haddad E, Puck JM, Kohn DB. Outcomes following treatment for ADA-deficient severe combined immunodeficiency: a report from the PIDTC. Blood. 2022 Aug 18;140(7):685-705. doi: 10.1182/blood.2022016196. PMID 35671392
- [Derived] Dorsey MJ, Wright NAM, Chaimowitz NS, Davila Saldana BJ, Miller H, Keller MD, Thakar MS, Shah AJ, Abu-Arja R, Andolina J, Aquino V, Barnum JL, Bednarski JJ, Bhatia M, Bonilla FA, Butte MJ, Bunin NJ, Chandra S, Chaudhury S, Chen K, Chong H, Cuvelier GDE, Dalal J, DeFelice ML, DeSantes KB, Forbes LR, Gillio A, Goldman F, Joshi AY, Kapoor N, Knutsen AP, Kobrynski L, Lieberman JA, Leiding JW, Oshrine B, Patel KP, Prockop S, Quigg TC, Quinones R, Schultz KR, Seroogy C, Shyr D, Siegel S, Smith AR, Torgerson TR, Vander Lugt MT, Yu LC, Cowan MJ, Buckley RH, Dvorak CC, Griffith LM, Haddad E, Kohn DB, Logan B, Notarangelo LD, Pai SY, Puck J, Pulsipher MA, Heimall J. Infections in Infants with SCID: Isolation, Infection Screening, and Prophylaxis in PIDTC Centers. J Clin Immunol. 2021 Jan;41(1):38-50. doi: 10.1007/s10875-020-00865-9. Epub 2020 Oct 2. PMID 33006109
- [Derived] Heimall J, Logan BR, Cowan MJ, Notarangelo LD, Griffith LM, Puck JM, Kohn DB, Pulsipher MA, Parikh S, Martinez C, Kapoor N, O'Reilly R, Boyer M, Pai SY, Goldman F, Burroughs L, Chandra S, Kletzel M, Thakar M, Connelly J, Cuvelier G, Davila Saldana BJ, Shereck E, Knutsen A, Sullivan KE, DeSantes K, Gillio A, Haddad E, Petrovic A, Quigg T, Smith AR, Stenger E, Yin Z, Shearer WT, Fleisher T, Buckley RH, Dvorak CC. Immune reconstitution and survival of 100 SCID patients post-hematopoietic cell transplant: a PIDTC natural history study. Blood. 2017 Dec 21;130(25):2718-2727. doi: 10.1182/blood-2017-05-781849. Epub 2017 Oct 11. PMID 29021228
- See also: Primary Immune Deficiency Treatment Consortium (PIDTC) featured highlights — https://www.rarediseasesnetwork.org/spotlight/v9i1/PIDTC
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Rare Diseases Clinical Research Network (RDCRN) — https://www.rarediseasesnetwork.org/cms/pidtc
- See also: National Center for Advancing Translational Science (NCATS) — https://ncats.nih.gov/